CLINICAL TRIAL: NCT00982813
Title: Prospective Study of the Influence of Periodontal Diseases on Pre-term Birth: Observation in the Maternity Hospital of Nantes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of internal organization
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BRD 09/4-G
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Periodontal Disease
Keywords: Periodontal disease; Per-term delivery; Sulcular bleeding index; Bacteriological gingival presence; Cytokines; Active periodontal disease with sulcular bleeding index; Bacteriological sampling in periodontal pocketing; Cytokines in the periodontal pocketing
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Periodontal screening — Periodontal screening in all patients giving birth between 24 and 37 gestational weeks.
  Bacteriological sampling in the periodontal pocketing. Search for specific cytokines in the periodontal pocketing. Professional prophylaxis and oral hygiene instruction.

SUMMARY:
The aim of the study is to determine the influence of the periodontal diseases in patients giving pre-term birth in the maternity hospital of Nantes. A French population is observed. The clinical, bacteriological and microbiological aspects will confirmed a comparative study which aim is dental prevention in the beginning of the pregnancy to avoid premature delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18
* Pre-term birth between 24 and 37 gestational weeks

Exclusion Criteria:

* Patient's opposition
* Delivery before 24 gestational weeks or after 37 gestational weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sulcular bleeding index as active disease | one week after delivery

SECONDARY OUTCOMES:
Plaque index | one week after delivery
Depth of periodontal pocketing | one week after delivery
Clinical attachment level | one week after delivery
Bacterial sampling of gingival crevicular fluid | One week after delivery
Search for cytokines in the gingival crevicular fluid | one week after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Henri-Jean PHILIPPE, Prof., Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France